CLINICAL TRIAL: NCT05703204
Title: A Phase 1 Clinical Study on the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of QLF32101 in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: A Study of QLF32101 in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLF32101-101
Record Dates: First submitted 2023-01-11; First posted 2023-01-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia and Myelodysplastic Syndrome
MeSH Terms: conditions — GATA2 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLF32101 (Experimental): single arm with QLF32101 treatment
  Interventions: Drug: QLF32101

INTERVENTIONS:
Drug: QLF32101 — The dose is given weekly and observed for 28 days(DLT observation period).Single agent treatment.

SUMMARY:
This study aimed to evaluate the safety,tolerability and preliminary efficacy of QLF32101 administered intravenously and subcutaneously in patients with R/R, AML.

DETAILED DESCRIPTION:
This open label, first-in-human study consists of 2 parts. Part 1 consists of dose escalation cohorts and Part 2 is expansion cohort.

The study population will include adult AML patients with relapse or refractory disease. In addition, in Part 2 medium and high-risk MDS patients are eligible.

In Part 1, dose escalations cohorts are followed until dose-limiting toxicity (DLT) or a maximum tolerated dose (MTD) or RecommendedPart2Dose (RP2D) is defined. Dose escalation decisions will be made by the Data Review Committee and will be primarily guided by safety data observed through the end of Cycle 1, as well as on-going assessment of safety beyond Cycle 1 in later cohorts.

Part 2 will begin once the MTD or RP2D is determined in Part 1. Part 2 will further characterize the safety, tolerability, Pharmacokinetic (PK), Pharmacodynamic (PD), immunogenicity and to assess preliminary efficacy of QLF32101.

ELIGIBILITY:
Inclusion Criteria:

1. Gender unlimited, age ≥ 18 years old;
2. Volunteer to participate in clinical trials and sign informed consent;
3. AML and medium-high risk MDS patients confirmed by histology and cytology;
4. Estimated survival time is at least 12 weeks;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2;
6. Any adverse event related to previous anti-tumor treatment must have returned to ≤ grade 1(NCI-CTCAE v5.0);
7. Main organ function is basically normal;
8. All female and male patients with reproductive ability must agree to take effective contraceptive methods during the study and within 6 months after the last use of the trial drug,the blood pregnancy test of female patients of childbearing age must be negative within 7 days before the first use of the study drug.

Exclusion Criteria:

1. Previously received hematopoietic stem cell transplantation;
2. Previous exposure to any anti-CLL-1 monoclonal antibody or CAR-T cell therapy;
3. Use other intervention study drugs within 4 weeks before the first use of the drug;
4. Any anti-tumor treatment received within 4 weeks before the first use of the drug;
5. Plan to vaccinate live attenuated vaccine within 4 weeks before the first use of the drug or during the study period;
6. Have received systemic glucocorticoid or other immunosuppressive therapy within 14 days before the first use of the drug;
7. With known central nervous system (CNS) leukemia infiltration;
8. ECG examination during screening period showed that QTcF>450 ms for males and 470 ms for females;
9. Major organ surgery within 4 weeks before the first use of the drug;
10. Received radiotherapy within 4 weeks before the first use of the drug;
11. There is an active infectious disease with clinical significance, which needs intravenous antibiotic treatment, and the investigator and sponsor judge that the patient is not suitable to participate in the clinical trial;
12. Chronic or acute active hepatitis B virus or hepatitis C virus infection;
13. Known active tuberculosis or active syphilis;
14. Known history of human immunodeficiency virus (HIV) infection；
15. Have received immunotherapy and have ≥ grade 3 immune related adverse events (irAE);
16. History of serious cardiovascular and cerebrovascular diseases;
17. History of other malignant tumors within 5 years before enrollment;
18. Breastfeeding patients；
19. Patients with known prior hypersensitivity to human or humanized monoclonal antibodies, or hypersensitivity to any of the components of QLF32101；
20. Have uncontrollable concomitant diseases or other diseases judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-08-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 28 Days
Maximum tolerated dose(MTD) | 28 Days
Recommended Phase II Dose (RP2D) | through study completion, an average of 1 year
R/R AML: cCR rate; Medium and high risk MDS: ORR (CR+complete remission of bone marrow [mCR]+PR+hematological improvement [HI]). | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Safety index:TEAEs,TRAEs,SAERs,TRSAEs. | through study completion, an average of 1 year
PK parameter | through study completion, an average of 1 year
Serum titer of ADAs against QLF32101 | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology&Blood Diseases Hospital,Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China